CLINICAL TRIAL: NCT03690271
Title: Study Programmed Intermittent Epidural Bolus (PIEB) vs PIEB: the Dose is it Variable According to the Patients
Brief Title: Study PIEB vs PIEB: the Dose is it Variable According to the Patients
Acronym: DOPABIEB
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3083_DOPABIEB
Record Dates: First submitted 2018-09-21; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia, Epidural; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Groupe 5-5: Patients for whom the clinician has prescribed local anesthetics in the epidural:
  * fixed dose administered every hour in a systematic way : 5 ml
  * dose to be administered every hour by the patient : 5 ml
- groupe 6-6: Patients for whom the clinician has prescribed local anesthetics in the epidural:
  * fixed dose administered every hour in a systematic way : 6 ml
  * dose to be administered every hour by the patient : 6 ml
- groupe 7-7: Patients for whom the clinician has prescribed local anesthetics in the epidural:
  * fixed dose administered every hour in a systematic way :7 ml
  * dose to be administered every hour by the patient :7 ml

SUMMARY:
the main objective of this study is to compare the effectiveness of three groups of epidurals with three different programmed intermittent epidural bolus (PIEB)settings.

DETAILED DESCRIPTION:
In a PIEB, the concentration of local anesthetics administered is standardized in the services according to the recommendations. What is left to the judgement of the clinician, taking care of the patient during the work, is the administered dose. This often varies according to clinician deductions that take notice of height, weight, previous pregnancies In the CHU of Rennes, three dosages are used in common practice. The objective by comparing these three dosages is to show if there is a significant difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Pregnant patient, during labor, live fetus, for whom a PIEB is desired / programmed.
* Patient not objecting to their participation in the study.

Exclusion Criteria:

* Hemostasis disorder contraindicated the epidural
* Eclampsia
* Caesarean section straightaway
* Patient under legal protection (guardianship, curatorship, safeguard of justice).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant patient, during labor, for whom a PIEB is desired / programmed.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
number of additional injections during work. | two days after infclusion

CONTACTS AND LOCATIONS:
Overall Officials: Eric WODEY, MD, PHD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France